CLINICAL TRIAL: NCT04024007
Title: Determination of Citrate Clearance Used in Regional Anticoagulation of Continuous Venous Hemofiltration Circuits
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr David DE BELS (Other)
Responsible Party: Sponsor-Investigator, Dr David DE BELS, Head of intensive care unit, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-citrate
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dialysis patients: Intensive care dialysis patients (Continuous Venous Hemofiltration with citrate). Dialysis performed according to the standard indications of the service. Patients are dialysed with the prismaflex system on AN69ST membranes.
  Interventions: Diagnostic Test: Citrate dosage

INTERVENTIONS:
Diagnostic Test: Citrate dosage — Patients are dialysed according to the standard of care. Biological variables are measured in pre-filter, post-filter and dialysate 30 minutes after the dialysis is initiated.

SUMMARY:
Citrate anticoagulation is becoming the gold standard in dialysis in intensive care units. It is now accepted that citrate prolongs the life of filters with a lower risk of bleeding.

However, the management of citrate is complex. Optimization is based on citrate flow, blood flow and the amount of calcium reinjected. Frequently the citrate level is sub-dosed.Currently, the fraction of excretion of citrate by the hemodialysis machine is unknown. Knowing this information would allow, if it is important enough, to add an additional parameter of citrate management by adapting the level of dialysis.

The determination of citrate in an extracorporeal circulation circuit has already been performed and has been validated in the literature. We propose to perform the assay on subjects with the same starting parameters, in order to deduce the clearance of citrate.

ELIGIBILITY:
Inclusion Criteria:

- Intensive care dialysis patients (Continuous Venous Hemofiltration with citrate).

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care dialysis patients (Continuous Venous Hemofiltration with citrate). Dialysis performed according to the standard indications of the service. Patients are dialysed with the prismaflex system on AN69ST membranes.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Citrate concentration - pre-filter | 30 minutes after the start of dialysis
  Citrate concentration in a blood sample taken before the dialysis filter
Citrate concentration - post-filter | 30 minutes after the start of dialysis
  Citrate concentration in a blood sample taken after the dialysis filter
Citrate concentration - dialysate | 30 minutes after the start of dialysis
  Citrate concentration in a blood sample taken in the dialysate

SECONDARY OUTCOMES:
Age | Baseline
  Age
Weight | Baseline
  Weight
Height | Baseline
  Height
Sex | Baseline
  Sex
Apache II score | Baseline
  The APACHE II score is calculated at the beginning of the intensive care unit admission to help determine the patient's mortality risk for the admission. An integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death.
SOFA (Sequential Organ Failure Assessment) score | Baseline
  The Sequential Organ Failure Assessment score (SOFA score), is used in intensive care units to determine and track the status of a patient with organ failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Higher scores mean a higher risk of mortality.
Glomerular filtration rate (GFR) | Baseline
  Glomerular filtration rate
Creatinin level | Baseline
  Creatinin level
Diuresis | Baseline
  Volume of urinary secretion in the last 12 hours
KDIGO classification | Baseline
  The KDIGO classification defines 3 stages of increasing severity for acute kidney injuries.
Na (sodium) concentration -pre-filter | 30 minutes after the start of dialysis
  Na (sodium) concentration in a blood sample taken before the dialysis filter
Na (sodium) concentration -post-filter | 30 minutes after the start of dialysis
  Na (sodium) concentration in a blood sample taken after the dialysis filter
Cl (chlorine) concentration - pre-filter | 30 minutes after the start of dialysis
  Cl (chlorine) concentration in a blood sample taken before the dialysis filter
Cl (chlorine) concentration -post-filter | 30 minutes after the start of dialysis
  Cl (chlorine) concentration in a blood sample taken after the dialysis filter
K (potassium) concentration - pre-filter | 30 minutes after the start of dialysis
  K (potassium) concentration in a blood sample taken before the dialysis filter
K (potassium) concentration - post-filter | 30 minutes after the start of dialysis
  K (potassium) concentration in a blood sample taken after the dialysis filter
Total Ca (calcium) concentration -pre-filter | 30 minutes after the start of dialysis
  Ca (calcium) concentration in a blood sample taken before the dialysis filter
Total Ca (calcium) concentration -post-filter | 30 minutes after the start of dialysis
  Ca (calcium) concentration in a blood sample taken after the dialysis filter
Total Ca (calcium) concentration -dialysate | 30 minutes after the start of dialysis
  Ca (calcium) concentration in the dialysate
Ionized calcium (Ca2+) concentration -pre-filter | 30 minutes after the start of dialysis
  Ca (calcium) concentration in a blood sample taken before the dialysis filter
Ionized calcium (Ca2+) concentration -post-filter | 30 minutes after the start of dialysis
  Ca (calcium) concentration in a blood sample taken after the dialysis filter
Ionized calcium (Ca2+) concentration -dialysate | 30 minutes after the start of dialysis
  Ca (calcium) concentration in the dialysate
Mg (magnesium) concentration - pre-filter | 30 minutes after the start of dialysis
  Mg (magnesium) concentration in a blood sample taken before the dialysis filter
Mg (magnesium) concentration - post-filter | 30 minutes after the start of dialysis
  Mg (magnesium) concentration in a blood sample taken after the dialysis filter
PO4 (phosphate) concentration - pre-filter | 30 minutes after the start of dialysis
  PO4 (phosphate) concentration in a blood sample taken before the dialysis filter
PO4 (phosphate) concentration - post-filter | 30 minutes after the start of dialysis
  PO4 (phosphate) concentration in a blood sample taken after the dialysis filter
Lactate concentration - pre-filter | 30 minutes after the start of dialysis
  Lactate blood concentration in a blood sample taken before the dialysis filter
Lactate concentration - post-filter | 30 minutes after the start of dialysis
  Lactate blood concentration in a blood sample taken after the dialysis filter
Albumin concentration -pre-filter | 30 minutes after the start of dialysis
  Albumin concentration in a blood sample taken before the dialysis filter
Albumin concentration -post-filter | 30 minutes after the start of dialysis
  Albumin concentration in a blood sample taken after the dialysis filter
pH - pre-filter | 30 minutes after the start of dialysis
  pH of a blood sample taken before the dialysis filter
pH - post-filter | 30 minutes after the start of dialysis
  pH of a blood sample taken after the dialysis filter
Total C-reactive protein (CRP) -pre-filter | 30 minutes after the start of dialysis
  Total CRP concentration in a blood sample taken before the dialysis filter
Total C-reactive protein (CRP) -post-filter | 30 minutes after the start of dialysis
  Total CRP concentration in a blood sample taken after the dialysis filter
Total C-reactive protein (CRP) -dialysate | 30 minutes after the start of dialysis
  Total CRP concentration in a blood sample taken in the dialysate
Monomeric C-reactive protein (CRP) -pre-filter | 30 minutes after the start of dialysis
  Monomeric CRP concentration in a blood sample taken before the dialysis filter
Monomeric C-reactive protein (CRP) -post-filter | 30 minutes after the start of dialysis
  Monomeric CRP concentration in a blood sample taken after the dialysis filter
Monomeric C-reactive protein (CRP) -dialysate | 30 minutes after the start of dialysis
  Monomeric CRP concentration in a blood sample taken in the dialysate

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Redant, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No